CLINICAL TRIAL: NCT03276273
Title: The Utility of Using the Bispectral Index (BIS) for Detecting Dialysis Disequilibrium Syndrome (DDS)
Brief Title: Bispectral-Electroencephalography (EEG) in First Time Hemodialysis
Acronym: BIS7
Status: Recruiting | Type: Observational
Sponsor: Suez Canal University (Other)
Collaborators: Dalian Medical University (Other)
Responsible Party: Principal Investigator, Ashraf A. Dahaba, Principal Investigator, Suez Canal University
Other Study IDs: MUGraz7
Record Dates: First submitted 2017-09-02; First posted 2017-09-08 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Renal Failure Acute Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: recording of Bispectral Index — recording of Bispectral Index

SUMMARY:
The severity of minimal dialysis disequilibrium syndrome (DDS) is currently detected and graded clinically using clinical criteria. Bispectral Index (BIS), an electroencephalographic (EEG) derived parameter is widely used in anesthesia and Critical Care setting to detect effects of anesthetic/hypnotic drugs. The aim of our study was to assess the discriminative power of BIS monitoring to accurately detect DDS.

DETAILED DESCRIPTION:
Design: A consecutive, clinical, validation study. Setting: Medical University of Graz (Graz, Austria). Patients: Twenty consecutive patients undergoing first hemodialysis are enrolled at Medical University of Graz, Haemodialysis Unit. Agitated patients or patients who fell asleep during the recording are excluded from the final analysis.

During the first dialysis session of approximately 3 h, patients were observed for signs of disequilibrium; headaches, dizziness, nausea, vomiting, if they become obtunded, have visual impairments or cramps. Accordingly patients were divided into 2 groups; the "DDS group" of patients who experienced one of the DDS symptoms of headaches, dizziness, nausea, vomiting, become obtunded, have visual impairments or cramps and patients who do not experience any of the DDS symptoms in the "non-DDS group" An assigned nephrologist will assess the physical and mental status of the patients.

ELIGIBILITY:
Inclusion Criteria:

* First Time renal Dialysis

Exclusion Criteria:

* subjects' consumption of sedatives/hypnotics psychotropic drugs, or concomitant neurological disorders affecting mental state such as hepatic encephalopathy, stroke, stupor or dementia and renal transplant patients.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First Time renal Dialysis
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Bispectral Index value | Over a period of one year Time point 1= First Hemodialysis, Time point 2= Second Hemodialysis, Time point 3= Third Hemodialysis.
  Interpatient Change in the value of recorded Bispectral Index between patients undergoing first time hemodialysis (differences between patients) and intrapatient (differences in bispectral Index values between the first 3 hemodialysis sections of each recruited patient)

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Dahaba, MD, Principal Investigator — Guest Professor
Locations (2):
- Dalian Medical University, Dalian, China
- Theodor Bilharz Research Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No